CLINICAL TRIAL: NCT05978076
Title: Serum Lipase and Severity of Pancreatic Injury.
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN472021/CHUSTE
Record Dates: First submitted 2023-07-25; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Injury
Keywords: Lipase; Pancreatic trauma; Pseudocysts
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Every children with elevated serum lipase: Every children with elevated serum lipase after trauma during those years will be included.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection : mechanism of injury, associated injury, length of stay, maximal lipase level, nutritional care and local complications.

SUMMARY:
Diagnosis of pancreas injury is not easy at first consult. It's a retrospective study, in children under 15 years and 3months, between January 1st 2010 to August 31th 2019, to prove that the first level of lipase is correlated with the severity of pancreatic injury.

Every children with elevated serum lipase after trauma during those years will be selected.

The children with pancreatic tumors will be excluded. American Association of Surgeon Trauma (AAST) classification of pancreas injury will be used to grade severity.

Children will be divided in two groups : one including pancreatic lesion with duct injury and one without duct injury.

Data will include mechanism of injury, associated injury, length of stay, maximal lipase level, nutritional care and local complications will be noted.

DETAILED DESCRIPTION:
The main objective of this study is to determine if there is a correlation between the initial serum lipase and the severity of the pancreatic injury.

ELIGIBILITY:
Inclusion Criteria:

* Children under 15 years 3 months with elevated lipase serum level after trauma.

Exclusion Criteria:

* Elevation of lipase secondary to pancreatic tumor

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 15 years 3 months with elevated lipase serum level after trauma will be included.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
lipase level in severe pancreatic injury (duct injury) | Month: 9 (end of study)
  Collected in medical history.
lipase level in light pancreatic injury (without duct injury) | Month: 9 (end of study)
  Collected in medical history.

SECONDARY OUTCOMES:
Local complications | Month: 9 (end of study)
  Collected in medical history.
Maximal lipase level | Month: 9 (end of study)
  Collected in medical history.

CONTACTS AND LOCATIONS:
Overall Officials: Aurélien SCALABRE, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- CHU Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No